CLINICAL TRIAL: NCT01940887
Title: A Phase 3 Randomized, Double-masked, Controlled Trial to Establish the Safety and Efficacy of Intravitreous Administration of Fovista® (Anti PDGF-B Pegylated Aptamer) Administered in Combination With Either Avastin® or Eylea® Compared to Avastin® or Eylea® Monotherapy in Subjects With Subfoveal Neovascular Age-related Macular Degeneration.
Brief Title: A Phase 3 Safety and Efficacy Study of Fovista® (E10030) Intravitreous Administration in Combination With Either Avastin® or Eylea® Compared to Avastin® or Eylea® Monotherapy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Ophthotech Corporation (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPH1004
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Results first posted 2020-09-30 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2020-09

CONDITIONS: Age-Related Macular Degeneration
Keywords: Wet AMD; choroidal neovascularization; Fovista®; E10030; Avastin®; Eylea®
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — E10030 aptamer; Bevacizumab; aflibercept; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- E10030 + bevacizumab or aflibercept (Experimental): E10030 1.5 mg intravitreal injection + bevacizumab 1.25 mg intravitreal injection or aflibercept 2 mg intravitreal injection
  Interventions: Drug: E10030; Drug: bevacizumab or aflibercept
- Sham + bevacizumab or aflibercept (Active Comparator): E10030 sham injection + bevacizumab 1.25 mg intravitreal injection or aflibercept 2 mg intravitreal injection
  Interventions: Drug: bevacizumab or aflibercept; Drug: E10030 sham injection

INTERVENTIONS:
Drug: E10030
  Other Names: Fovista®
  Arms: E10030 + bevacizumab or aflibercept
Drug: bevacizumab or aflibercept — Patients are randomized to receive either bevacizumab or aflibercept
  Other Names: Avastin®; Eylea®
Drug: E10030 sham injection — Pressure on the eye with a syringe with no needle
  Other Names: Sham
  Arms: Sham + bevacizumab or aflibercept

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of intravitreal administration of Fovista® administered in combination with either Avastin® or Eylea® compared to Avastin® or Eylea® monotherapy in subjects with subfoveal choroidal neovascularization secondary to age-related macular degeneration (AMD).

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1 ratio to the following two arms per study design:

* Fovista® 1.5 mg/eye + Avastin® 1.25 mg/eye or Eylea® 2 mg/eye
* Fovista® sham + Avastin® 1.25 mg/eye or Eylea® 2 mg/eye

Subjects will be treated for up to 24 months with active Fovista® or sham, in combination with either Avastin® or Eylea® with the primary endpoint at 12 months.

Approximately 622 subjects will be randomized into one of the two treatment groups (311 patients per dose group), and the efficacy analysis will be based on the data from these two groups as per the SAP

ELIGIBILITY:
Inclusion Criteria:

* Subjects of either gender aged ≥ 50 years
* Active subfoveal choroidal neovascularization (CNV) secondary to AMD
* Presence of sub-retinal hyper-reflective material (SD-OCT)

Exclusion Criteria:

* Any prior treatment for AMD in the study eye prior to the Day 1 visit, except oral supplements of vitamins and minerals
* Any prior intravitreal treatment in the study eye prior to the Day 1 visit, regardless of indication (including intravitreal corticosteroids)
* Any intraocular surgery or thermal laser within three (3) months of trial entry. Any prior thermal laser in the macular region, regardless of indication
* Subjects with subfoveal scar or subfoveal atrophy are excluded
* Diabetes mellitus

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (174):
- United States (91):
  - Gilbert, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Campbell, California
  - Fresno, California
  - Fullerton, California
  - Irvine, California
  - La Jolla, California
  - Mountain View, California
  - Palm Desert, California
  - Redlands, California
  - Sacramento, California
  - San Francisco, California
  - Santa Ana, California
  - Ventura, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Golden, Colorado
  - Hamden, Connecticut
  - New London, Connecticut
  - Altamonte Springs, Florida
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Largo, Florida
  - Melbourne, Florida
  - Palm Beach Gardens, Florida
  - Pensacola, Florida
  - St. Petersburg, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Marietta, Georgia
  - Oak Forest, Illinois
  - Peoria, Illinois
  - West Des Moines, Iowa
  - Leawood, Kansas
  - Shawnee Mission, Kansas
  - Topeka, Kansas
  - Wichita, Kansas
  - Paducah, Kentucky
  - Baltimore, Maryland
  - Chevy Chase, Maryland
  - Hagerstown, Maryland
  - Towson, Maryland
  - Boston, Massachusetts
  - Peabody, Massachusetts
  - Worcester, Massachusetts
  - Jackson, Michigan
  - Lansing, Michigan
  - Southfield, Michigan
  - Minneapolis, Minnesota
  - Chesterfield, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Reno, Nevada
  - Lawrenceville, New Jersey
  - Albuquerque, New Mexico
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - Asheville, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Camp Hill, Pennsylvania
  - Philadelphia, Pennsylvania
  - West Mifflin, Pennsylvania
  - Ladson, South Carolina
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Abilene, Texas
  - Amarillo, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - McAllen, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Willow Park, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Bellevue, Washington
  - Silverdale, Washington
  - Morgantown, West Virginia
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Santa Fe
- Australia (5):
  - Albury, New South Wales
  - Parramatta, New South Wales
  - Sydney, New South Wales
  - Westmead, New South Wales
  - East Melbourne, Victoria
- Graz, Austria
- Brazil (2):
  - Goiânia
  - São Paulo
- Canada (4):
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Mississauga, Ontario
  - Montral, Quebec
- Colombia (2):
  - Bogotá
  - Medellín
- Croatia (3):
  - Osijek
  - Rijeka
  - Zagreb
- Czechia (4):
  - Brno
  - Hradec Králové
  - Olomouc
  - Prague
- Tallinn, Estonia
- Finland (2):
  - Helsinki
  - Kuopio
- France (7):
  - Créteil
  - Lyon
  - Marseille
  - Paris
  - Rouen
  - Strasbourg
  - Tours
- Germany (10):
  - Münster, Norhdhein-Westfalen
  - Aachen, North Rhine-Westphalia
  - Leipzig, Saxony
  - Kiel, Schleswig-Holstein
  - Göttingen
  - Hamburg
  - Karlsruhe
  - Lübeck
  - Mainz
  - Tübingen
- Hungary (5):
  - Budapest
  - Debrecen
  - Pécs
  - Szeged
  - Veszprém
- Israel (6):
  - Haifa
  - Jerusalem
  - Kfar Saba
  - Pita Tikva
  - Rehovot
  - Tel Aviv
- Italy (8):
  - Ancona
  - Bologna
  - Ferrara
  - Milan
  - Padua
  - Roma
  - Torino
  - Udine
- Riga, Latvia
- Stavanger, Norway
- Poland (4):
  - Bydgoszcz
  - Katowice
  - Lodz
  - Wroclaw
- Portugal (4):
  - Coimbra
  - Lisbon
  - Porto
  - Vila Franca de Xira
- Slovakia (2):
  - Banská Bystrica
  - Trenčín
- Spain (8):
  - Las Palmas de Gran Canaria, Canary Islands
  - Pamplona, Navarre
  - Bilbao, Vizcaya
  - A Coruña
  - Albacete
  - Barcelona
  - Oviedo
  - Valencia

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 214 centers (107 in North America and 107 in the rest of the world) in 22 countries (20 of which enrolled patients) between 19 May 2014 and 15 September 2017.
Pre-assignment Details: Three (3) of the 645 patients who were enrolled and randomized did not receive treatments. Remaining 642 subjects were grouped into two treatment groups (E10030 + Eylea/Avastin vs. Sham + Eylea/Avastin) for the purposes of efficacy analyses in accordance with the pre-specified study design, and the SAP.
Groups:
- E10030 + Bevacizumab or Aflibercept: E10030 1.5 mg intravitreal injection + bevacizumab 1.25 mg intravitreal injection or aflibercept 2 mg intravitreal injection
  E10030
  bevacizumab or aflibercept: Patients are randomized to receive either bevacizumab or aflibercept
Period: Year 1
Arm/Group | E10030 + Bevacizumab or Aflibercept | Sham + Bevacizumab or Aflibercept
Started | 322 | 320
Completed | 283 | 297
Not Completed | 39 | 23
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 7 | 3
Not completed — Death | 5 | 3
Not completed — Adverse Event | 7 | 6
Not completed — Withdrawal by Subject | 18 | 9
Not completed — Lost to Follow-up | 2 | 1
Period: Year 2
Arm/Group | E10030 + Bevacizumab or Aflibercept | Sham + Bevacizumab or Aflibercept
Started | 283 | 297
Completed | 66 | 75
Not Completed | 217 | 222
Not completed — Physician Decision | 8 | 1
Not completed — Death | 0 | 2
Not completed — Sponsor Decision, early termination | 192 | 203
Not completed — Adverse Event | 8 | 2
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Lost to Follow-up | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E10030 + Bevacizumab or Aflibercept | Sham + Bevacizumab or Aflibercept | Total
Number analyzed (Participants) | 322 | 320 | 642
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.5 (8.36) | 76.6 (8.36) | 76.6 (8.36)
Age, Customized [Count of Participants; unit: Participants]
  Age: Adults 18-64 years | 31 | 25 | 56
  Age: Adults 65-84 years | 239 | 239 | 478
  Age: Adults 85 years and over | 52 | 56 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 192 | 370
  Male | 144 | 128 | 272
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 23 | 51
  Not Hispanic or Latino | 294 | 297 | 591
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Colombia | 7 | 5 | 12
  Argentina | 4 | 4 | 8
  Hungary | 48 | 50 | 98
  United States | 92 | 95 | 187
  Czechia | 15 | 14 | 29
  Portugal | 9 | 12 | 21
  Spain | 10 | 10 | 20
  Canada | 1 | 1 | 2
  Austria | 2 | 3 | 5
  Latvia | 8 | 7 | 15
  Poland | 1 | 3 | 4
  Brazil | 3 | 3 | 6
  Italy | 28 | 29 | 57
  Israel | 32 | 28 | 60
  Slovakia | 1 | 0 | 1
  Australia | 2 | 3 | 5
  France | 26 | 23 | 49
  Croatia | 22 | 21 | 43
  Estonia | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Acuity (Measured at Baseline and at the Month 12 Visit)
Description: The primary efficacy endpoint is the mean change in visual acuity (ETDRS letters) measured at baseline and at the month 12 visit. Higher ETDRS letters represents higher vision and a higher change in ETDRS letters represents better functioning.
Time Frame: 12 months
Population: As pre-specified in the SAP and per the study design, 2 treatment groups (E10030 +Eylea/Avastin vs. Sham + Eylea/Avastin) will be compared. All 642 subjects who received at least one dose of the study drug, irrespective of the dose received, were included in the analysis.
Measure: Mean (Standard Error); unit: letters
Arm/Group | E10030 + Bevacizumab or Aflibercept | Sham + Bevacizumab or Aflibercept
Number analyzed (Participants) | 322 | 320
letters | 9.42 (0.85) | 9.04 (0.85)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality data was collected for up to 2 years, and Adverse events (AEs) were collected for up to 12 months of exposure (Year 1) for the 2 pre-specified treatment groups (E10030 + Bevacizumab or Aflibercept vs. Sham + Bevacizumab or Aflibercept), per the study design and the SAP.
Description: AEs in the safety population (all subjects who received at least one dose of the study treatment) were collected for up to 12 months of exposure (Year 1). All AEs that ultimately resulted in death (regardless of the actual date of death) were included in All Cause Mortality count, and hence the count may differ from the Participant Flow Table which included reported deaths at the time of early discontinuation from the study.
Arm/Group | E10030 + Bevacizumab or Aflibercept | Sham + Bevacizumab or Aflibercept
All-Cause Mortality (participants affected / at risk) | 7/322 | 6/320
Serious Adverse Events (participants affected / at risk) | 58/322 | 32/320
Other Adverse Events (participants affected / at risk) | 105/322 | 107/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E10030 + Bevacizumab or Aflibercept (N=322) | Sham + Bevacizumab or Aflibercept (N=320)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 3 (3)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Autoimmune uveitis (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Corneal endotheliitis (Eye disorders) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (2) | 1 (2)
Retinal haemorrhage (Eye disorders) | 2 (3) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric dysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Device dislocation (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 4 (4) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Nosocomial infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (2)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E10030 + Bevacizumab or Aflibercept (N=322) | Sham + Bevacizumab or Aflibercept (N=320)
Intraocular pressure increased (Investigations) | 22 (46) | 20 (35)
Conjunctival haemorrhage (Eye disorders) | 39 (85) | 31 (48)
Punctate keratitis (Eye disorders) | 21 (34) | 14 (39)
Eye pain (Eye disorders) | 18 (26) | 21 (35)
Vitreous detachment (Eye disorders) | 20 (21) | 19 (23)
Neovascular age-related macular degeneration (Eye disorders) | 16 (16) | 19 (19)
Nasopharyngitis (Infections and infestations) | 14 (15) | 17 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution agrees not to individually publish the results of the Study without Ophthotech's prior written consent. Institution may participate in a joint, multi-center publications of the Study results with the other investigators and/or institutions only, upon prior written consent of Ophthotech.

DOCUMENTS (2):
  • Study Protocol (2014-03-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT01940887/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT01940887/SAP_001.pdf